CLINICAL TRIAL: NCT03523728
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Two Stage Study to Characterize the Efficacy, Safety, Tolerability and Pharmacokinetics of GZ/SAR402671 in Patients at Risk of Rapidly Progressive Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: A Medical Research Study Designed to Determine if Venglustat Can be a Future Treatment for ADPKD Patients
Acronym: STAGED-PKD
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Interim analysis for futility of the Stage 1 of the EFC15392 study met the protocol specified stopping rule based on the primary endpoint. EFC15392 study was stopped for futility based on prespecified criteria and recommendation from DMC
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC15392; 2017-004084-12 (EudraCT Number); U1111-1202-0775 (Other: UTN)
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Results first posted 2022-11-09 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — venglustat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Stage 1- Placebo (Placebo Comparator): Participants from Stage 1 were randomized to receive 2 capsules of placebo matched to venglustat once daily for treatment period of 24 months.
  Interventions: Drug: Placebo
- Stage 1- Venglustat 8 mg (Experimental): Participants from Stage 1 were randomized to receive venglustat 8 milligrams (mg) (i.e., 2 capsules of 4 mg) once daily for treatment period of 24 months.
  Interventions: Drug: Venglustat
- Stage 1- Venglustat 15 mg (Experimental): Participants from Stage 1 were randomized to receive 1 capsule of venglustat 15 mg and 1 capsule of placebo matched to venglustat once daily for treatment period of 24 months.
  Interventions: Drug: Venglustat; Drug: Placebo
- Stage 2- Placebo (Placebo Comparator): Participants from Stage 2 were randomized to receive 1 capsule of placebo matched to venglustat once daily for treatment period of 24 months.
  Interventions: Drug: Placebo
- Stage 2- Venglustat 15 mg (Experimental): Participants from Stage 2 were randomized to receive 1 capsule of venglustat 15 mg once daily for treatment period of 24 months.
  Interventions: Drug: Venglustat

INTERVENTIONS:
Drug: Venglustat — Pharmaceutical form: capsule; Route of administration: oral
  Other Names: GZ402671
  Arms: Stage 1- Venglustat 15 mg; Stage 1- Venglustat 8 mg; Stage 2- Venglustat 15 mg
Drug: Placebo — Pharmaceutical form: capsule; Route of administration: oral
  Arms: Stage 1- Placebo; Stage 1- Venglustat 15 mg; Stage 2- Placebo

SUMMARY:
Primary Objective:

To determine the effect of venglustat on the rate of total kidney volume (TKV) growth (Stage 1) and estimated glomerular filtration rate (eGFR) decline in participants at risk of rapidly progressive Autosomal Dominant Polycystic Kidney Disease (ADPKD) (Stage 2).

Secondary Objectives:

* To determine the effect of venglustat on the rate of renal function decline (Stage 1) and on the rate of TKV growth (Stage 2).
* To evaluate the pharmacokinetics (PK) of venglustat in ADPKD participants (Stages 1 and 2).
* To determine the effect of venglustat on pain and fatigue, based on participant reported diary (Stages 1 and 2).
* Safety/tolerability objectives:
* To characterize the safety profile of venglustat (Stages 1 and 2).
* To evaluate the effect of venglustat on mood using Beck Depression Inventory II (BDI-II) (Stages 1 and 2).
* To evaluate the effect of venglustat on the lens by ophthalmological examination (Stages 1 and 2).

DETAILED DESCRIPTION:
Study duration per participant was 26 months (maximal) that included a screening period of 15 days, run-in period of 2 weeks, a 24-month treatment period, and a follow-up 30 days after final dose of investigational medicinal product (IMP).

ELIGIBILITY:
Inclusion criteria:

* Male or female adult with ADPKD with age at the time the consent was signed:

  1. between 18 to 50 years (both inclusive) for participants from Stage 1.
  2. between 18 to 50 years (both inclusive) for participants from Stage 2 with eGFR between 45 and 89.9 milliliters per minute per 1.73 meter square (mL/min/1.73 m^2) during screening period.*
  3. between 18 to 55 years (both inclusive) for participants from Stage 2 with eGFR between 30 and 44.9 mL/min/1.73 m^2 during screening period.*
* Diagnosis of ADPKD in participants with a family history would be based on unified Pei criteria. In the absence of a family history, the diagnosis would be based on the presence of renal cysts bilaterally, totaling at least 20, in the absence of findings suggestive of other cystic renal diseases.
* Mayo Imaging Classification of ADPKD Class 1C, 1D or 1E**

  **Total kidney volume (TKV) had confirmed by a central reader prior to Visit 3.
* Estimated glomerular filtration rate between 45 to 89.9 mL/min/1.73 m^2 during screening period* (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation) for Stage 1.
* Estimated glomerular filtration rate between 30 to 89.9 mL/min/1.73 m^2 during screening period* (CKD-EPI equation) for Stage 2.

  *Eligibility would be confirmed by eGFR value from one of the two first pre-randomization eGFR measurements.
* Stable treatment regimen of antihypertensive therapy for at least 30 days prior to the screening visit for hypertensive participant.
* Able to read, comprehend, and respond to the study questionnaires.
* Participant had given voluntary written informed consent before performance of any study related procedures not part of standard medical care.
* Participant had no access to tolvaptan at the time of study start or tolvaptan was not indicated for treatment of participant according to treating physician (participant does not meet recommended criteria for treatment, refuses to initiate or does not tolerate treatment with tolvaptan).
* The participants, if female of childbearing potential, must have had a negative blood pregnancy test (β-human chorionic gonadotropin [β-hCG]) at the screening visit and a negative urine pregnancy test at the baseline visit.
* Female participants of childbearing potential and male participants must have had agreed to practice true abstinence in line with their preferred and usual lifestyle or to use double-contraceptive methods (including a highly effective method of contraception for female participants of childbearing potential) for the entire duration of the study and for at least 6 weeks for females and 90 days for males following their last dose of study drug.

Exclusion criteria:

* Systolic blood pressure greater than (>) 160 millimeters of Mercury (mmHg) at Run-in and Baseline visits.
* Administration within 3 months prior to the screening visit of tolvaptan or other Polycystic Kidney Disease-modifying agents (somatostatin analogues).
* Participation in another investigational interventional study or use of IMP, within 3 months or 5 half lives, whichever was longer, before randomization.
* The participant had a positive result of any of the following tests: hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (anti HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti HIV1 and anti HIV2 Ab). Participants with a positive hepatitis B surface antibody (HBsAb) test were eligible if other criteria were met (i.e., negative tests for: HBsAg, hepatitis B core antibody [HBcAb]). Participants immune due to natural infection (positive hepatitis B surface antibody (HBsAb), negative hepatitis B surface antigen (HBsAg) and positive hepatitis B core antibody [HBcAb]) were eligible if they had negative hepatitis B vaccine (HBV) deoxyribonucleic acid (DNA) test.
* A history of drug and/or alcohol abuse within the past year prior to the screening visit. A history of alcohol dependence within the 5 years prior to the screening visit.
* The participant was scheduled for in-patient hospitalization including elective surgery, during the study.
* The participant had a clinically significant, uncontrolled medical condition that, in the opinion of the investigator, would put the safety of the participant at risk through participation, or which would affect the efficacy or safety analysis if the condition exacerbated during the study, or that might significantly interfere with study compliance, including all prescribed evaluations and follow-up activities.
* The participants, in the opinion of the investigator, was unable to adhere to the requirements of the study or unable to undergo study assessments (e.g., had contraindications to pupillary dilation or unable to undergo magnetic resonance imaging (MRI) [For example: participant's weight exceeds weight capacity of the MRI, ferromagnetic metal prostheses, aneurysm clips, severe claustrophobia, large abdominal/back tattoos, etc.]).
* Any country-related specific regulation that would prevent the participant from entering the study.
* The participants did not adhere to treatment (less than [<] 70 percent [%] compliance rate) in the run-in.
* The participant had, according to World Health Organization (WHO) Grading, a cortical cataract greater than or equal to (>=)one-quarter of the lens circumference (Grade cortical cataract-2 [COR-2]) or a posterior subcapsular cataract >=2 millimeter (Grade posterior subcapsular cataract-2 [PSC-2]). Participant with nuclear cataracts would not be excluded.
* The participant was then receiving potentially cataractogenic medications, including a chronic regimen (more frequently than every 2 weeks) of any route of corticosteroids (including medium and high potency topical steroids) or any medication that might cause cataract, according to the Prescribing Information.
* The participant had received strong or moderate inducers or inhibitors of CYP3A4 within 14 days or 5 half-lives, whichever was longer, prior to randomization. This also included the consumption of grapefruit, grapefruit juice, or grapefruit containing products within 72 hours of starting venglustat administration.
* The participant was pregnant, or lactating.
* Liver enzymes (alanine aminotransferase /aspartate aminotransferase ) or total bilirubin >2 times the upper limit of normal unless the participant had the diagnosis of Gilbert syndrome. Participants with the Gilbert syndrome should have had no additional symptoms or signs which suggested hepatobiliary disease and serum total bilirubin level no more than 3 milligrams per deciliter (mg/dL) (51 [micromoles per Liter] mcmol/L) with conjugated bilirubin less than 20% of the total bilirubin fraction.
* Presence of severe depression as measured by Beck Depression Inventory-II (BDI-II) >28 and/or a history of a major affective disorder within 1 year of the screening visit.
* Known hypersensitivity to venglustat or any component of the excipients.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 478 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (95):
- United States (18):
  - Investigational Site Number 8400002, Birmingham, Alabama
  - Investigational Site Number 8400017, Los Angeles, California
  - Investigational Site Number 8400001, San Francisco, California
  - Investigational Site Number 8400008, Aurora, Colorado
  - Investigational Site Number 8400010, New Haven, Connecticut
  - Investigational Site Number 8400004, Atlanta, Georgia
  - Investigational Site Number 8400007, Chicago, Illinois
  - Investigational Site Number 8400014, Iowa City, Iowa
  - Investigational Site Number 8400003, Kansas City, Kansas
  - Investigational Site Number 8400021, Baltimore, Maryland
  - Investigational Site Number 8400016, Boston, Massachusetts
  - Investigational Site Number 8400020, Rochester, Minnesota
  - Investigational Site Number 8400027, Kansas City, Missouri
  - Investigational Site Number 8400011, Philadelphia, Pennsylvania
  - Investigational Site Number 8400015, San Antonio, Texas
  - Investigational Site Number 8400019, Morgantown, West Virginia
  - Investigational Site Number 8400005, Madison, Wisconsin
  - Investigational Site Number 8400006, Milwaukee, Wisconsin
- Argentina (2):
  - Investigational Site Number 0320001, Buenos Aires
  - Investigational Site Number 0320003, Santa Fe
- Australia (3):
  - Investigational Site Number 0360002, Herston
  - Investigational Site Number 0360003, Nedlands
  - Investigational Site Number 0360001, Westmead
- Austria (2):
  - Investigational Site Number 0400001, Graz
  - Investigational Site Number 0400004, Vienna
- Belgium (2):
  - Investigational Site Number 0560001, Brussels
  - Investigational Site Number 0560002, Leuven
- Canada (3):
  - Investigational Site Number 1240002, Edmonton
  - Investigational Site Number 1240003, Montreal
  - Investigational Site Number 1240001, Toronto
- China (9):
  - Investigational Site Number 1560005, Beijing
  - Investigational Site Number 1560004, Chengdu
  - Investigational Site Number 1560009, Guangzhou
  - Investigational Site Number 1560006, Hangzhou
  - Investigational Site Number 1560002, Hefei
  - Investigational Site Number 1560007, Nanjing
  - Investigational Site Number 1560008, Nanjing
  - Investigational Site Number 1560001, Shanghai
  - Investigational Site Number 1560003, Shenyang
- Czechia (2):
  - Investigational Site Number 2030001, Prague
  - Investigational Site Number 2030002, Prague
- Denmark (2):
  - Investigational Site Number 2080001, Copenhagen
  - Investigational Site Number 2080002, Roskilde
- France (4):
  - Investigational Site Number 2500004, Bordeaux
  - Investigational Site Number 2500003, Brest
  - Investigational Site Number 2500002, Paris
  - Investigational Site Number 2500001, Toulouse
- Germany (10):
  - Investigational Site Number 2760001, Berlin
  - Investigational Site Number 2760003, Cologne
  - Investigational Site Number 2760002, Dresden
  - Investigational Site Number 2760010, Dresden
  - Investigational Site Number 2760007, Düsseldorf
  - Investigational Site Number 2760009, Essen
  - Investigational Site Number 2760005, Hanover
  - Investigational Site Number 2760011, Leipzig
  - Investigational Site Number 2760012, Mainz
  - Investigational Site Number 2760004, München
- Israel (2):
  - Investigational Site Number 3760003, Ashdod
  - Investigational Site Number 3760002, Rehovot
- Italy (3):
  - Investigational Site Number 3800001, Brescia
  - Investigational Site Number 3800002, Milan
  - Investigational Site Number 3800003, Napoli
- Japan (10):
  - Investigational Site Number 3920002, Bunkyō City
  - Investigational Site Number 3920005, Kamakura-Shi
  - Investigational Site Number 3920006, Kawasaki-Shi
  - Investigational Site Number 3920010, Kyoto
  - Investigational Site Number 3920009, Nagoya
  - Investigational Site Number 3920003, Niigata
  - Investigational Site Number 3920007, Osaka
  - Investigational Site Number 3920001, Sapporo
  - Investigational Site Number 3920004, Shinjuku-Ku
  - Investigational Site Number 3920008, Toyoake-Shi
- Netherlands (3):
  - Investigational Site Number 5280003, Amsterdam
  - Investigational Site Number 5280001, Groningen
  - Investigational Site Number 5280002, Nijmegen
- Poland (3):
  - Investigational Site Number 6160001, Lodz
  - Investigational Site Number 6160003, Warsaw
  - Investigational Site Number 6160002, Wroclaw
- Portugal (3):
  - Investigational Site Number 6200004, Almada
  - Investigational Site Number 6200005, Carnaxide
  - Investigational Site Number 6200001, Loures
- Romania (3):
  - Investigational Site Number 6420002, Bucharest
  - Investigational Site Number 6420004, Oradea
  - Investigational Site Number 6420001, Timișoara
- South Korea (2):
  - Investigational Site Number 4100001, Seoul
  - Investigational Site Number 4100002, Seoul
- Spain (3):
  - Investigational Site Number 7240003, Barcelona
  - Investigational Site Number 7240001, Barcelona
  - Investigational Site Number 7240002, Madrid
- Taiwan (2):
  - Investigational Site Number 1580001, Taichung
  - Investigational Site Number 1580002, Taipei
- Turkey (Türkiye) (3):
  - Investigational Site Number 7920001, Istanbul
  - Investigational Site Number 7920002, Kayseri
  - Investigational Site Number 7920003, Kocaeli
- Investigational Site Number 8260001, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Gansevoort RT, Hariri A, Minini P, Ahn C, Chapman AB, Horie S, Knebelmann B, Mrug M, Ong ACM, Pei YPC, Torres VE, Modur V, Antonshchuk I, Perrone RD. Venglustat, a Novel Glucosylceramide Synthase Inhibitor, in Patients at Risk of Rapidly Progressing ADPKD: Primary Results of a Double-Blind, Placebo-Controlled, Phase 2/3 Randomized Clinical Trial. Am J Kidney Dis. 2023 May;81(5):517-527.e1. doi: 10.1053/j.ajkd.2022.10.016. Epub 2022 Dec 17. PMID 36535535
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Perrone RD, Hariri A, Minini P, Ahn C, Chapman AB, Horie S, Knebelmann B, Mrug M, Ong ACM, Pei YPC, Torres VE, Modur V, Gansevoort RT. The STAGED-PKD 2-Stage Adaptive Study With a Patient Enrichment Strategy and Treatment Effect Modeling for Improved Study Design Efficiency in Patients With ADPKD. Kidney Med. 2022 Aug 27;4(10):100538. doi: 10.1016/j.xkme.2022.100538. eCollection 2022 Oct. PMID 36204243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 93 sites that enrolled participants in 23 countries. A total of 478 participants were enrolled from 04 October 2018 to 01 June 2021. Study was conducted in 2 stages: Stage 1 and Stage 2.
Pre-assignment Details: Participants who completed 24 months of treatment in either Stage 1 or Stage 2 of EFC15392 had option to enroll in an open-label long-term extension study LTS15823 (NCT ID: NCT04705051).
Period: Stage 1 (24 Months)
Arm/Group | Stage 1- Placebo | Stage 1- Venglustat 8 mg | Stage 1- Venglustat 15 mg | Stage 2- Placebo | Stage 2- Venglustat 15 mg
Started | 78 | 78 | 80 | 0 | 0
Completed | 12 | 10 | 12 | 0 | 0
Not Completed | 66 | 68 | 68 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 4 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0
Not completed — Poor compliance to protocol | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 5 | 7 | 0 | 0
Not completed — Study terminated by sponsor | 54 | 59 | 56 | 0 | 0
Not completed — Other-Unspecified | 1 | 2 | 0 | 0 | 0
Period: Stage 2 (24 Months)
Arm/Group | Stage 1- Placebo | Stage 1- Venglustat 8 mg | Stage 1- Venglustat 15 mg | Stage 2- Placebo | Stage 2- Venglustat 15 mg
Started | 0 | 0 | 0 | 123 (Stage 1 and Stage 2 were separate population.) | 119 (Stage 1 and Stage 2 were separate population.)
Treated | 0 | 0 | 0 | 122 | 119
Estimated Glomerular Filtration Rate (eGFR) Between 45 and 89.9 mL/Min/1.73 m^2 at Screening | 0 | 0 | 0 | 97 | 90
eGFR Between 30 and 44.9 mL/Min/1.73 m^2 at Screening | 0 | 0 | 0 | 25 | 29
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 123 | 119
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 119 | 110
Not completed — Other-Unspecified | 0 | 0 | 0 | 2 | 3
Not completed — Randomized and not treated | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants randomized in the study.
Groups:
- Stage 1- Venglustat 8 mg: Participants from Stage 1 were randomized to receive venglustat 8 mg (i.e., 2 capsules of 4 mg) once daily for treatment period of 24 months.
Arm/Group | Stage 1- Placebo | Stage 1- Venglustat 8 mg | Stage 1- Venglustat 15 mg | Stage 2- Placebo | Stage 2- Venglustat 15 mg | Total Title
Number analyzed (Participants) | 78 | 78 | 80 | 123 | 119 | 478
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (6.0) | 41.7 (6.9) | 43.6 (5.7) | 41.7 (6.9) | 42.1 (6.7) | 42.2 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 31 | 34 | 46 | 48 | 196
  Male | 41 | 47 | 46 | 77 | 71 | 282
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 27 | 27 | 27 | 52 | 55 | 188
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 2 | 0 | 3
  White | 48 | 50 | 52 | 66 | 64 | 280
  More than one race | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 0 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Annualized Slope of Change in Total Kidney Volume (TKV) From Baseline to Month 18: Stage 1
Description: Total kidney volume is a measure for assessing disease progression in participants with ADPKD, a prognostic biomarker of renal function decline and progression to end-stage renal disease. Kidney volume was assessed using magnetic resonance imaging (MRI). The annualized slope of change in TKV (in percentage [%] per year) in each treatment group was obtained from the back-transformation of the mean slope of log10-transformed TKV obtained from the linear mixed effect model. The model included fix effects of treatment (venglustat 15 mg, venglustat 8 mg or placebo), mayo imaging classification (as per randomization stratification factor: class 1C versus 1D versus 1E), time (as continuous variable in years), treatment * time interaction and mayo imaging classification * time interaction and included random intercept and slope.
Time Frame: From Baseline to Month 18
Population: Analysis was performed on Stage 1 intent-to-treat (ITT) population that includes all participants randomized in Stage 1 and were analyzed according to the intervention allocated by randomization (venglustat 15 mg, venglustat 8 mg or placebo). Here, 'Overall number of participants analyzed' signifies participants who were evaluable for the outcome measure.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percent change in TKV/year
Arm/Group | Stage 1- Placebo | Stage 1- Venglustat 8 mg | Stage 1- Venglustat 15 mg
Number analyzed (Participants) | 78 | 78 | 79
percent change in TKV/year | 6.35 [5.10 to 7.62] | 7.71 [6.46 to 8.98] | 6.38 [5.11 to 7.66]
Statistical Analysis 1: Comparison: Stage 1- Placebo vs Stage 1- Venglustat 8 mg; Test type: Superiority; p = 0.1367, linear mixed effect model; Relative difference = 21.32, 95% CI 2-sided [-5.77 to 58.22]
Statistical Analysis 2: Comparison: Stage 1- Placebo vs Stage 1- Venglustat 15 mg; Test type: Superiority; p = 0.9812, linear mixed effect model; Relative difference = 0.34, 95% CI 2-sided [-24.57 to 33.36]

2. Primary Outcome: Annualized Rate of Change in Estimated Glomerular Filtration Rate (eGFR) (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) From Baseline to Month 24: Combined Stage 1 and Stage 2
Description: An eGFR was used to measure level of kidney function and determine the stage of kidney disease in ADPKD participants. Baseline eGFR was defined for each participant as the average of eGFR values assessed prior or equal to first dose of study drug or randomization for participants randomized and not exposed. Annualized rate of change in eGFR in each treatment group was obtained from the linear mixed effect model including the fixed categorical effects of treatment group (venglustat 15 mg, venglustat 8 mg or placebo), mayo imaging classification (as per interactive response technology [IRT]: 1C, 1D, 1E), time (as continuous variable in years), treatment-by-time, mayo imaging classification-by-time, and included random intercept and slope.
Time Frame: From Baseline to Month 24
Population: Analysis was performed on Combined Stage 1 and Stage 2 ITT population that included all participants with an eGFR between 45 and 89.9 mL/min/1.73 m^2 at screening who are randomized in Stage 1 or Stage 2 and were analyzed according to the intervention allocated by randomization (venglustat 15 mg, venglustat 8 mg or placebo). Data for this outcome measure (OM) was planned to be collected and analyzed for combined Stage 1 and Stage 2 population as pre-specified in protocol.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2/year
Groups:
- Placebo: All participants from Stage 1 or Stage 2 were randomized to receive placebo matched to venglustat once daily for treatment period of 24 months.
- Venglustat 8 mg: Participants from Stage 1 were randomized to receive venglustat 8 mg (i.e., 2 capsules of 4 mg) once daily for treatment period of 24 months.
- Venglustat 15 mg: All participants from Stage 1 or Stage 2 were randomized to receive 1 capsule of venglustat 15 mg once daily for treatment period of 24 months.
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 175 | 78 | 170
mL/min/1.73 m^2/year | -2.40 [-3.30 to -1.49] | -4.82 [-5.82 to -3.83] | -4.89 [-5.80 to -3.99]
Statistical Analysis 1: Comparison: Placebo vs Venglustat 8 mg; Test type: Superiority; p = 0.0005, linear mixed effect model; Relative difference = 101.32, 95% CI 2-sided [35.63 to 233.72]
Statistical Analysis 2: Comparison: Placebo vs Venglustat 15 mg; Test type: Superiority; p = 0.0002, linear mixed effect model; Relative difference = 104.17, 95% CI 2-sided [39.54 to 236.45]

3. Secondary Outcome: Annualized Rate of Change in Estimated Glomerular Filtration Rate (eGFR) From Baseline to Month 24: Stage 1
Description: An eGFR was used to measure level of kidney function and determine the stage of kidney disease in ADPKD participants. Baseline eGFR was defined for each participant as the average of eGFR values assessed prior or equal to first dose of study drug or randomization for participants randomized and not exposed. Annualized rate of change in eGFR was obtained from the linear mixed effect model including the fixed categorical effects of treatment group, mayo imaging classification (as per IRT), time (as continuous variable in years), treatment-by-time, mayo imaging classification-by-time, and included random intercept and slope. Due to early termination of study for futility, the two-steps analysis initially planned was not applicable, then the annualized rate of change from baseline in eGFR in Stage 1 population were assessed using all data available up to database lock (i.e., including Month 24 assessment). As this is a slope, it allowed to have more data and to reduce variability.
Time Frame: From Baseline to Month 24
Population: Analysis was performed on Stage 1 ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2/year
Arm/Group | Stage 1- Placebo | Stage 1- Venglustat 8 mg | Stage 1- Venglustat 15 mg
Number analyzed (Participants) | 78 | 78 | 80
mL/min/1.73 m^2/year | -3.14 [-4.09 to -2.18] | -4.74 [-5.68 to -3.80] | -4.59 [-5.53 to -3.65]
Statistical Analysis 1: Comparison: Stage 1- Placebo vs Stage 1- Venglustat 8 mg; Test type: Superiority; p = 0.0197, linear mixed effect model; Relative difference = 51.01, 95% CI 2-sided [7.01 to 125.45]
Statistical Analysis 2: Comparison: Stage 1- Placebo vs Stage 1- Venglustat 15 mg; Test type: Superiority; p = 0.0337, linear mixed effect model; Relative difference = 46.36, 95% CI 2-sided [3.21 to 119.01]

4. Secondary Outcome: Annualized Slope of Change in Total Kidney Volume (TKV) From Baseline to Month 18: Combined Stage 1 and Stage 2
Description: Total kidney volume is a measure for assessing disease progression in participants with ADPKD, a prognostic biomarker of renal function decline and progression to end-stage renal disease. Kidney volume was assessed using MRI. The annualized slope of change in TKV (in % per year) in each treatment group was obtained from the back-transformation of the mean slope of log10-transformed TKV obtained from the linear mixed effect model. The model included fix effects of treatment (venglustat 15 mg, venglustat 8 mg or placebo), mayo imaging classification (as per randomization stratification factor: class 1C versus 1D versus 1E), time (as continuous variable in years), treatment * time interaction and mayo imaging classification * time interaction and included random intercept and slope.
Time Frame: From Baseline to Month 18
Population: As no post-baseline MRI data were collected in Stage 2 due to early study discontinuation, the analysis of TKV in Combined Stage 1 and Stage 2 was not done.
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change in Pain Severity as Measured by Brief Pain Inventory-Short Form (BPI-SF)-Item 3 Scale Score From Baseline to Month 18: Stage 1
Description: The BPI-SF is a validated, self-administered questionnaire designed to measure a participant's perceived level of pain. The BPI-SF consisted of 15 items that use a numeric rating scale (NRS) to assess pain severity and pain interference in the past 24 hours and the past week. BPI-SF Item 3 asks participants to "Please rate your pain by marking the box beside the number that best describes your pain at its worst in the past 24 hours." The NRS ranged from 0 (no pain) to 10 (worst imaginable pain), where higher scores indicates greater intensity of pain. Least-squares (LS) means, and standard errors (SE) were estimated from mixed-effect model with repeated measures (MMRM) analysis.
Time Frame: From Baseline to Month 18
Population: Analysis was performed on Stage 1 ITT population. Here, 'Overall number of participants analyzed' signifies participants who were evaluable for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage 1- Placebo | Stage 1- Venglustat 8 mg | Stage 1- Venglustat 15 mg
Number analyzed (Participants) | 69 | 65 | 65
score on a scale | -0.09 (0.15) | 0.01 (0.17) | -0.35 (0.16)
Statistical Analysis 1: Comparison: Stage 1- Placebo vs Stage 1- Venglustat 8 mg; Test type: Superiority; p = 0.6374, Mixed effect model with repeated measure; Least square mean difference = 0.11, 95% CI 2-sided [-0.342 to 0.556], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Stage 1- Placebo vs Stage 1- Venglustat 15 mg; Test type: Superiority; p = 0.2560, Mixed effect model with repeated measure; Least square mean difference = -0.25, 95% CI 2-sided [-0.689 to 0.185], Standard Error of Mean 0.22

6. Secondary Outcome: Change in Pain Severity as Measured by Brief Pain Inventory-Short Form (BPI-SF)-Item 3 Scale Score From Baseline to Month 24: Combined Stage 1 and Stage 2
Description: The BPI-SF is a validated, self-administered questionnaire designed to measure a participant's perceived level of pain. The BPI-SF consisted of 15 items that use a NRS to assess pain severity and pain interference in the past 24 hours and the past week. BPI-SF Item 3 asks participants to "Please rate your pain by marking the box beside the number that best describes your pain at its worst in the past 24 hours." The NRS ranged from 0 (no pain) to 10 (worst imaginable pain), where higher scores indicate greater intensity of pain. LS means and SE were estimated from MMRM analysis.
Time Frame: From Baseline to Month 24
Population: Analysis was performed on Combined Stage 1 and Stage 2 ITT population. Here, 'Overall number of participants analyzed' signifies participants who were evaluable for the outcome measure. Data for this OM was planned to be collected and analyzed for combined Stage 1 and Stage 2 population as pre-specified in protocol.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 133 | 65 | 126
score on a scale | -0.20 (0.23) | -0.31 (0.36) | -0.36 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Venglustat 8 mg; Test type: Superiority; p = 0.7900, Mixed effect model with repeated measure; Least square mean difference = -0.11, 95% CI 2-sided [-0.971 to 0.747], Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: Placebo vs Venglustat 15 mg; Test type: Superiority; p = 0.6322, Mixed effect model with repeated measure; Least square mean difference = -0.15, 95% CI 2-sided [-0.808 to 0.500], Standard Error of Mean 0.32

7. Secondary Outcome: Change in Fatigue Severity as Measured by Brief Fatigue Inventory (BFI-SF)-Item 3 Scale Score From Baseline to Month 18: Stage 1
Description: The BFI-SF is a 10-item, validated, self-administered questionnaire that was originally developed to assess fatigue severity. The 10-items were measured on a 0-10 scale, with 0 being 'does not interfere' and 10 being 'completely interferes.' BFI - Item 3 asks participants to 'Please rate your fatigue (weariness, tiredness) by circling the one number that best describes your worst level of fatigue during the past 24 hours. The NRS ranged from 0 (no fatigue) to 10 (worst imaginable fatigue). Higher global scores were associated with more severe fatigue. LS means and SE were estimated from MMRM analysis.
Time Frame: From Baseline to Month 18
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Stage I- Venglustat 15 mg: Participants from Stage 1 were randomized to receive 1 capsule of venglustat 15 mg and 1 capsule of placebo matched to venglustat once daily for treatment period of 24 months.
Arm/Group | Stage 1- Placebo | Stage 1- Venglustat 8 mg | Stage I- Venglustat 15 mg
Number analyzed (Participants) | 69 | 65 | 65
score on a scale | -0.26 (0.23) | -0.10 (0.25) | -0.64 (0.24)
Statistical Analysis 1: Comparison: Stage 1- Placebo vs Stage 1- Venglustat 8 mg; Test type: Superiority; p = 0.6245, Mixed effect model with repeated measure; Least square mean difference = 0.17, 95% CI 2-sided [-0.506 to 0.839], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Stage 1- Placebo vs Stage I- Venglustat 15 mg; Test type: Superiority; p = 0.2567, Mixed effect model with repeated measure; Least square mean difference = -0.38, 95% CI 2-sided [-1.044 to 0.281], Standard Error of Mean 0.33

8. Secondary Outcome: Change in Fatigue Severity as Measured by Brief Fatigue Inventory (BFI-SF)-Item 3 Scale Score From Baseline to Month 24: Combined Stage 1 and Stage 2
Description: The BFI-SF is a 10-item, validated, self-administered questionnaire that was originally developed to assess fatigue severity. The 10-items were measured on a 0-10 scale, with 0 being 'does not interfere' and 10 being 'completely interferes.' BFI - Item 3 asks participants to "Please rate your fatigue (weariness, tiredness) by circling the one number that best describes your worst level of fatigue during the past 24 hours. The NRS ranged from 0 (no fatigue) to 10 (worst imaginable fatigue). Higher global scores were associated with more severe fatigue. LS means and SE were estimated from MMRM analysis.
Time Frame: From Baseline to Month 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 133 | 65 | 126
score on a scale | 0.02 (0.38) | -0.85 (0.55) | -0.51 (0.38)
Statistical Analysis 1: Comparison: Placebo vs Venglustat 8 mg; Test type: Superiority; p = 0.2023, Mixed effect model with repeated measure; Least square mean difference = -0.87, 95% CI 2-sided [-2.232 to 0.485], Standard Error of Mean 0.68
Statistical Analysis 2: Comparison: Placebo vs Venglustat 15 mg; Test type: Superiority; p = 0.3205, Mixed effect model with repeated measure; Least square mean difference = -0.54, 95% CI 2-sided [-1.610 to 0.537], Standard Error of Mean 0.53

9. Secondary Outcome: Pharmacokinetics: Plasma Concentration of Venglustat: Stage 1
Description: Venglustat plasma concentrations was determined using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method. Data for this outcome measure was not planned to be collected and analyzed for placebo arm.
Time Frame: Day 1: 3 hours Post-Dose, Month 1: Pre-Dose and 3 hours Post-Dose, Month 6: Pre-Dose, Month 18: Pre-Dose
Population: Analysed on Stage 1 pharmacokinetic (PK) population that included all participants randomized in Stage 1 who took at least one dose of study drug and had at least one post-baseline PK assessment; analyzed according to the intervention they actually received. Here, "number analyzed" signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Stage 1- Venglustat 8 mg | Stage 1- Venglustat 15 mg
Number analyzed (Participants) | 78 | 80
nanograms per milliliter
  Day 1: 3 hours Post-Dose: number analyzed (Participants) | 65 | 73
  Day 1: 3 hours Post-Dose | 27.8 (11.9) | 50.9 (22.5)
  Month 1: Pre-Dose: number analyzed (Participants) | 72 | 63
  Month 1: Pre-Dose | 54.7 (19.2) | 103.9 (50.2)
  Month 1: 3 hours Post-Dose: number analyzed (Participants) | 75 | 64
  Month 1: 3 hours Post-Dose | 82.1 (24.7) | 154.6 (61.1)
  Months 6: Pre-Dose: number analyzed (Participants) | 47 | 54
  Months 6: Pre-Dose | 57.5 (23.5) | 106.2 (56.3)
  Months 18: Pre-Dose: number analyzed (Participants) | 41 | 41
  Months 18: Pre-Dose | 58.3 (22.0) | 120.3 (73.1)

10. Secondary Outcome: Pharmacokinetics: Plasma Concentration of Venglustat: Stage 2
Description: Venglustat plasma concentrations was determined using a validated LC-MS/MS method. Data for this outcome measure was not planned to be collected and analyzed for placebo arm.
Time Frame: Month 1: Pre-dose and 3 hours Post-dose
Population: Analysis was performed on Stage 2 PK population that included all participants with an eGFR between 45 and 89.9 mL/min/1.73 m^2 at screening who were randomized in Stage 2, who took at least one dose of study drug and who had at least one post-baseline PK assessment. Participants were analyzed according to study drug they actually received. Here, "number analyzed" signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Stage 2- Venglustat 15 mg
Number analyzed (Participants) | 77
nanograms per milliliter
  Month 1: Pre-Dose: number analyzed (Participants) | 60
  Month 1: Pre-Dose | 109.3 (60.7)
  Month 1: 3 hours Post-Dose: number analyzed (Participants) | 61
  Month 1: 3 hours Post-Dose | 163.5 (79.7)

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs): Stage 1
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. A serious adverse event (SAE) was any untoward medical occurrence that at any dose: results in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was a medically important event. TEAEs were AEs that developed, worsened or became serious during the treatment-emergent (TE) period (defined as the time from the first investigational medicinal product [IMP] administration up to the last IMP administration in EFC15392 study + 30 days or up to the first visit in LTS15823 study, whichever comes earlier).
Time Frame: From the first IMP administration up to the last IMP administration in EFC15392 study + 30 days (i.e., up to 25 months) or up to the first visit in LTS15823 study, whichever comes earlier
Population: Analysis was performed on Stage 1 safety population that included all participants randomized in Stage 1 who took at least one dose or part of a dose of the double-blind IMP, analyzed according to the treatment actually received (venglustat 15 mg, venglustat 8 mg, or placebo)
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1- Placebo | Stage 1- Venglustat 8 mg | Stage 1- Venglustat 15 mg
Number analyzed (Participants) | 78 | 78 | 80
Participants
  TEAEs | 62 | 65 | 70
  TESAEs | 8 | 15 | 19

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs): Combined Stage 1 and Stage 2
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. SAE was any untoward medical occurrence that at any dose: results in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was a medically important event. TEAEs were AEs that developed, worsened or became serious during the TE period (defined as the time from the first IMP administration up to the last IMP administration in EFC15392 study + 30 days or up to the first visit in LTS15823 study, whichever comes earlier).
Time Frame: as for outcome 11
Population: Analysis was performed on extended Combined Stage 1 and Stage 2 safety population that included all participants with an eGFR between 45 and 89.9 mL/min/1.73 m^2 at screening who were randomized in Stage 1 or Stage 2 and who took at least one dose or part of a dose of IMP, analyzed according to treatment actually received. Data for this OM was planned to be collected and analyzed for combined Stage 1 and Stage 2 population as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 200 | 78 | 199
Participants
  TEAEs | 128 | 65 | 143
  TESAEs | 14 | 15 | 26

13. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities: Hematology: Combined Stage 1 and Stage 2
Description: Criteria for potentially clinically significant abnormalities: Hemoglobin: less than or equal to (<=) 115 grams per liter (g/L) [Male]; <=95 g/L [Female]; greater than or equal to (>=) 185 g/L [Male]; >=165 g/L [Female]; Decrease from baseline >=20 g/L; Hematocrit: <=0.37 volume/volume (v/v) [Male]; <=0.32 v/v [Female]; >=0.55 v/v [Male]; >=0.5 v/v [Female]; Erythrocyte (red blood cells [RBC]): >=6*10^12 per liter (/L); Platelet: less than (<) 100*10^9/L; >=700*10^9/L; Leukocyte (white blood cells [WBC]): <3*10^9/L [Non-Black]; <2*10^9/L [Black], >=16*10^9/L; Neutrophils: <1.5*10^9/L [Non-Black]; <1*10^9/L [Black]; Lymphocytes: greater than (>) 4*10^9/L, Monocytes: >0.7*10^9/L; Basophils: >0.1*10^9/L; and Eosinophils: >0.5*10^9/L or >upper limit of normal (ULN) (if ULN >=0.5*10^9/L).
Time Frame: as for outcome 11
Population: Analysis was performed on extended Combined Stage 1 and Stage 2 safety population. Here, "number analyzed" signifies participants with available data for specified category. Data for this OM was planned to be collected and analyzed for combined Stage 1 and Stage 2 population as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 200 | 78 | 199
Participants
  Hemoglobin: <=115 g/L (Male); <=95 g/L (Female): number analyzed (Participants) | 187 | 78 | 190
  Hemoglobin: <=115 g/L (Male); <=95 g/L (Female) | 7 | 3 | 5
  Hemoglobin: >=185 g/L (Male); >=165 g/L (Female): number analyzed (Participants) | 187 | 78 | 190
  Hemoglobin: >=185 g/L (Male); >=165 g/L (Female) | 0 | 0 | 0
  Hemoglobin: Decrease from baseline >=20 g/L: number analyzed (Participants) | 186 | 78 | 190
  Hemoglobin: Decrease from baseline >=20 g/L | 4 | 7 | 5
  Hematocrit: <=0.37 v/v (Male); <=0.32 v/v (Female): number analyzed (Participants) | 186 | 78 | 190
  Hematocrit: <=0.37 v/v (Male); <=0.32 v/v (Female) | 40 | 20 | 42
  Hematocrit: >=0.55 v/v (Male); >=0.5 v/v (Female): number analyzed (Participants) | 186 | 78 | 190
  Hematocrit: >=0.55 v/v (Male); >=0.5 v/v (Female) | 0 | 0 | 0
  Erythrocyte (RBC): >=6 * 10^12/L: number analyzed (Participants) | 187 | 78 | 190
  Erythrocyte (RBC): >=6 * 10^12/L | 1 | 0 | 1
  Platelet: <100*10^9/L: number analyzed (Participants) | 187 | 78 | 190
  Platelet: <100*10^9/L | 0 | 2 | 1
  Platelet: >=700*10^9/L: number analyzed (Participants) | 187 | 78 | 190
  Platelet: >=700*10^9/L | 0 | 0 | 0
  Leukocyte (WBC): <3*10^9/L (Non-Black); <2*10^9/L (Black): number analyzed (Participants) | 187 | 78 | 190
  Leukocyte (WBC): <3*10^9/L (Non-Black); <2*10^9/L (Black) | 1 | 2 | 4
  Leukocyte (WBC): >=16*10^9/L: number analyzed (Participants) | 187 | 78 | 190
  Leukocyte (WBC): >=16*10^9/L | 0 | 2 | 1
  Neutrophils: <1.5*10^9/L (Non-Black); <1*10^9/L (Black): number analyzed (Participants) | 187 | 78 | 190
  Neutrophils: <1.5*10^9/L (Non-Black); <1*10^9/L (Black) | 1 | 1 | 3
  Lymphocytes: >4*10^9/L: number analyzed (Participants) | 187 | 78 | 190
  Lymphocytes: >4*10^9/L | 0 | 1 | 0
  Monocytes >0.7*10^9/L: number analyzed (Participants) | 187 | 78 | 190
  Monocytes >0.7*10^9/L | 6 | 3 | 7
  Basophils: >0.1*10^9/L: number analyzed (Participants) | 187 | 78 | 190
  Basophils: >0.1*10^9/L | 33 | 5 | 8
  Eosinophils: >0.5*10^9/L or >ULN: number analyzed (Participants) | 187 | 78 | 190
  Eosinophils: >0.5*10^9/L or >ULN | 7 | 2 | 1

14. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities: Clinical Chemistry: Combined Stage 1 and Stage 2
Description: Criteria for potentially clinically significant abnormalities: Glucose: <=3.9 millimoles per liter (mmol/L) and <lower limit of normal (LLN): >=11.1 mmol/L (unfasted); >=7 mmol/L (fasted); Albumin:<=25 g/L; Sodium: <=129 mmol/L; >=160 mmol/L; Potassium: <3 mmol/L; >=5.5 mmol/L; Chloride: <80 mmol/L, >115 mmol/L; Creatinine: >=150 micro millimoles per liter (mcmol/L) (Adults); >=30% change from Baseline; >=100% change from Baseline, Urea Nitrogen: >=17 mmol/L; Alanine Aminotransferase (ALT): >3 ULN; Aspartate Aminotransferase (AST): >3 ULN; Alkaline Phosphatase: >1.5 ULN; Total Bilirubin: >1.5 ULN, >2 ULN; ALT >3 ULN and Bilirubin >2 ULN; and Direct Bilirubin >35% Bilirubin and Bilirubin >1.5 ULN.
Time Frame: as for outcome 11
Population: Analysis was performed on extended Combined Stage 1 and Stage 2 safety population. Here, "number analyzed" signifies participants with available data for each specified category. Data for this OM was planned to be collected and analyzed for combined Stage 1 and Stage 2 population as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 200 | 78 | 199
Participants
  Glucose: <=3.9 mmol/L and <LLN: number analyzed (Participants) | 196 | 78 | 196
  Glucose: <=3.9 mmol/L and <LLN | 17 | 5 | 12
  Glucose: >=11.1 mmol/L (unfasted); >=7 mmol/L (fasted): number analyzed (Participants) | 196 | 78 | 196
  Glucose: >=11.1 mmol/L (unfasted); >=7 mmol/L (fasted) | 10 | 5 | 19
  Albumin: <=25 g/L: number analyzed (Participants) | 196 | 78 | 196
  Albumin: <=25 g/L | 0 | 0 | 0
  Sodium: <=129 mmol/L: number analyzed (Participants) | 196 | 78 | 196
  Sodium: <=129 mmol/L | 1 | 0 | 3
  Sodium: >=160 mmol/L: number analyzed (Participants) | 196 | 78 | 196
  Sodium: >=160 mmol/L | 0 | 0 | 0
  Potassium: <3 mmol/L: number analyzed (Participants) | 196 | 78 | 196
  Potassium: <3 mmol/L | 0 | 1 | 0
  Potassium: >=5.5 mmol/L: number analyzed (Participants) | 196 | 78 | 196
  Potassium: >=5.5 mmol/L | 5 | 5 | 11
  Chloride: <80 mmol/L: number analyzed (Participants) | 196 | 78 | 196
  Chloride: <80 mmol/L | 0 | 1 | 0
  Chloride: >115 mmol/L: number analyzed (Participants) | 196 | 78 | 196
  Chloride: >115 mmol/L | 1 | 0 | 0
  Creatinine: >=150 mcmol/L (Adults): number analyzed (Participants) | 196 | 78 | 196
  Creatinine: >=150 mcmol/L (Adults) | 50 | 21 | 70
  Creatinine: >=30% change from Baseline: number analyzed (Participants) | 196 | 78 | 196
  Creatinine: >=30% change from Baseline | 12 | 18 | 25
  Creatinine: >=100% change from Baseline: number analyzed (Participants) | 196 | 78 | 196
  Creatinine: >=100% change from Baseline | 0 | 1 | 4
  Urea Nitrogen: >=17 mmol/L: number analyzed (Participants) | 196 | 78 | 196
  Urea Nitrogen: >=17 mmol/L | 1 | 0 | 6
  ALT: > 3 ULN: number analyzed (Participants) | 196 | 78 | 196
  ALT: > 3 ULN | 0 | 0 | 0
  AST: >3 ULN: number analyzed (Participants) | 196 | 78 | 196
  AST: >3 ULN | 0 | 0 | 0
  Alkaline Phosphatase: >1.5 ULN: number analyzed (Participants) | 196 | 78 | 196
  Alkaline Phosphatase: >1.5 ULN | 3 | 0 | 0
  Total Bilirubin: >1.5 ULN: number analyzed (Participants) | 196 | 78 | 196
  Total Bilirubin: >1.5 ULN | 2 | 0 | 1
  Total Bilirubin: >2 ULN: number analyzed (Participants) | 196 | 78 | 196
  Total Bilirubin: >2 ULN | 0 | 0 | 0
  ALT >3 ULN and Bilirubin >2 ULN: number analyzed (Participants) | 196 | 78 | 196
  ALT >3 ULN and Bilirubin >2 ULN | 0 | 0 | 0
  Direct Bilirubin >35% Bilirubin and Bilirubin >1.5 ULN: number analyzed (Participants) | 195 | 78 | 196
  Direct Bilirubin >35% Bilirubin and Bilirubin >1.5 ULN | 2 | 0 | 0

15. Secondary Outcome: Number of Participants With Potentially and Clinically Significant Abnormalities: Urinalysis: Combined Stage 1 and Stage 2
Description: Criteria for potentially clinically significant abnormalities: Urine pH: <=4.6 and >=8.
Time Frame: as for outcome 11
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 200 | 78 | 199
Participants
  Urine pH: <=4.6: number analyzed (Participants) | 156 | 70 | 153
  Urine pH: <=4.6 | 0 | 0 | 0
  Urine pH: >=8: number analyzed (Participants) | 156 | 70 | 153
  Urine pH: >=8 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Potentially and Clinically Significant Abnormalities: Vital Signs: Combined Stage 1 and Stage 2
Description: Criteria for potentially clinically significant abnormalities: Sitting Systolic Blood Pressure: <=95 millimeters of Mercury (mmHg) and decrease from Baseline >=20 mmHg; >=160 mmHg and increase from Baseline >=20 mmHg; Sitting Diastolic Blood Pressure: <=45 mmHg and decrease from Baseline >=10 mmHg, >=110 mmHg and increase from Baseline >=10 mmHg; Sitting Heart Rate: <=50 beats/minute and decrease from Baseline >=20 beats/minute; >=120 beats/minute and increase from Baseline >=20 beats/minute; and Weight: >=5% decrease from Baseline; >=5% increase from Baseline.
Time Frame: as for outcome 11
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 200 | 78 | 199
Participants
  Sitting Systolic Blood Pressure: <=95 mmHg and decrease from Baseline >=20 mmHg: number analyzed (Participants) | 196 | 78 | 196
  Sitting Systolic Blood Pressure: <=95 mmHg and decrease from Baseline >=20 mmHg | 0 | 0 | 1
  Sitting Systolic Blood Pressure: >=160 mmHg and increase from Baseline >=20 mmHg: number analyzed (Participants) | 196 | 78 | 196
  Sitting Systolic Blood Pressure: >=160 mmHg and increase from Baseline >=20 mmHg | 2 | 3 | 10
  Sitting Diastolic Blood Pressure: <= 45 mmHg and decrease from Baseline >=10 mmHg: number analyzed (Participants) | 196 | 78 | 196
  Sitting Diastolic Blood Pressure: <= 45 mmHg and decrease from Baseline >=10 mmHg | 0 | 0 | 0
  Sitting Diastolic Blood Pressure: >=110 mmHg and increase from Baseline >=10 mmHg: number analyzed (Participants) | 196 | 78 | 196
  Sitting Diastolic Blood Pressure: >=110 mmHg and increase from Baseline >=10 mmHg | 2 | 4 | 7
  Sitting Heart Rate: <=50 beats/min and decrease from Baseline >=20 beats/min: number analyzed (Participants) | 196 | 78 | 196
  Sitting Heart Rate: <=50 beats/min and decrease from Baseline >=20 beats/min | 0 | 2 | 2
  Sitting Heart Rate: >=120 beats/min and increase from Baseline >=20 beats/min: number analyzed (Participants) | 196 | 78 | 196
  Sitting Heart Rate: >=120 beats/min and increase from Baseline >=20 beats/min | 0 | 0 | 0
  Weight: >=5% decrease from Baseline: number analyzed (Participants) | 156 | 70 | 155
  Weight: >=5% decrease from Baseline | 11 | 4 | 13
  Weight: >=5% increase from Baseline: number analyzed (Participants) | 156 | 70 | 155
  Weight: >=5% increase from Baseline | 15 | 9 | 15

17. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities: Electrocardiogram: Combined Stage 1 and Stage 2
Description: Criteria for potentially clinically significant abnormalities: Heart Rate: <50 beats/minute; <50 beats/minute and decrease from Baseline >=20 beats/minute; <40 beats/minute; <40 beats/minute and decrease from Baseline >=20 beats/min; <30 beats/minute; >90 beats/minute; >90 beats/minute and increase from Baseline >=20 beats/minute; >100 beats/minute; >100 beats/minute and increase from Baseline >=20 beats/minute; >120 beats/minute; >120 beats/minute, increase from Baseline >=20 beats/minute; PR Interval: >200 milliseconds (msec); >200 msec and increase from Baseline >=25%; >220 msec, >240 msec; QRS Interval: >110 msec; >110 msec and increase from Baseline >=25%; >120 msec; >120 msec and increase from Baseline >=25%; QT Interval: >500 msec; QT corrected for heart rate (QTc) Bazett: >450 msec; >480 msec; increase from Baseline (30-60) msec; increase from Baseline >60 msec; QTc Fridericia: >450 msec; >480 msec; increase from Baseline (30-60) msec and increase from Baseline > 60 msec.
Time Frame: as for outcome 11
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 200 | 78 | 199
Participants
  Heart Rate: <50 beats/min: number analyzed (Participants) | 140 | 70 | 132
  Heart Rate: <50 beats/min | 7 | 6 | 13
  Heart Rate: <50 beats/min and decrease from Baseline >=20 beats/min: number analyzed (Participants) | 140 | 70 | 132
  Heart Rate: <50 beats/min and decrease from Baseline >=20 beats/min | 1 | 0 | 1
  Heart Rate: <40 beats/min: number analyzed (Participants) | 140 | 70 | 132
  Heart Rate: <40 beats/min | 0 | 1 | 1
  Heart Rate: <40 beats/min and decrease from Baseline >=20 beats/min: number analyzed (Participants) | 140 | 70 | 132
  Heart Rate: <40 beats/min and decrease from Baseline >=20 beats/min | 0 | 0 | 0
  Heart Rate: <30 beats/min: number analyzed (Participants) | 140 | 70 | 132
  Heart Rate: <30 beats/min | 0 | 0 | 0
  Heart Rate: >90 beats/min: number analyzed (Participants) | 140 | 70 | 132
  Heart Rate: >90 beats/min | 4 | 2 | 3
  Heart Rate: >90 beats/min and increase from Baseline >=20 beats/min: number analyzed (Participants) | 140 | 70 | 132
  Heart Rate: >90 beats/min and increase from Baseline >=20 beats/min | 2 | 2 | 2
  Heart Rate: >100 beats/min: number analyzed (Participants) | 140 | 70 | 132
  Heart Rate: >100 beats/min | 1 | 0 | 2
  Heart Rate: >100 beats/min and increase from Baseline >=20 beats/min: number analyzed (Participants) | 140 | 70 | 132
  Heart Rate: >100 beats/min and increase from Baseline >=20 beats/min | 1 | 0 | 1
  Heart Rate: >120 beats/min: number analyzed (Participants) | 140 | 78 | 132
  Heart Rate: >120 beats/min | 0 | 0 | 0
  Heart Rate: >120 beats/min and increase from Baseline >=20 beats/min: number analyzed (Participants) | 140 | 70 | 132
  Heart Rate: >120 beats/min and increase from Baseline >=20 beats/min | 0 | 0 | 0
  PR Interval: >200 msec: number analyzed (Participants) | 140 | 70 | 132
  PR Interval: >200 msec | 8 | 2 | 10
  PR Interval: >200 msec and increase from Baseline >=25%: number analyzed (Participants) | 140 | 70 | 132
  PR Interval: >200 msec and increase from Baseline >=25% | 0 | 0 | 0
  PR Interval: >220 msec: number analyzed (Participants) | 140 | 70 | 132
  PR Interval: >220 msec | 1 | 0 | 2
  PR Interval: >240 msec: number analyzed (Participants) | 140 | 70 | 132
  PR Interval: >240 msec | 0 | 0 | 0
  QRS Interval: >110 msec: number analyzed (Participants) | 140 | 70 | 132
  QRS Interval: >110 msec | 11 | 4 | 10
  QRS Interval: > 110 msec and increase from Baseline >=25%: number analyzed (Participants) | 140 | 70 | 132
  QRS Interval: > 110 msec and increase from Baseline >=25% | 0 | 0 | 1
  QRS Interval: >120 msec: number analyzed (Participants) | 140 | 70 | 132
  QRS Interval: >120 msec | 2 | 1 | 3
  QRS Interval: >120 msec and increase from Baseline >=25%: number analyzed (Participants) | 140 | 70 | 132
  QRS Interval: >120 msec and increase from Baseline >=25% | 0 | 0 | 1
  QT Interval: >500 msec: number analyzed (Participants) | 140 | 70 | 132
  QT Interval: >500 msec | 0 | 0 | 0
  QTc Bazett: >450 msec: number analyzed (Participants) | 140 | 70 | 132
  QTc Bazett: >450 msec | 5 | 2 | 3
  QTc Bazett: >480 msec: number analyzed (Participants) | 140 | 70 | 132
  QTc Bazett: >480 msec | 0 | 0 | 0
  QTc Bazett: Increase from Baseline [30-60] msec: number analyzed (Participants) | 136 | 68 | 128
  QTc Bazett: Increase from Baseline [30-60] msec | 13 | 1 | 5
  QTc Bazett: Increase from Baseline >60 msec: number analyzed (Participants) | 136 | 68 | 128
  QTc Bazett: Increase from Baseline >60 msec | 0 | 0 | 0
  QTc Fridericia: >450 msec: number analyzed (Participants) | 140 | 70 | 132
  QTc Fridericia: >450 msec | 4 | 1 | 2
  QTc Fridericia: >480 msec: number analyzed (Participants) | 140 | 70 | 132
  QTc Fridericia: >480 msec | 0 | 0 | 0
  QTc Fridericia: Increase from Baseline [30-60] msec: number analyzed (Participants) | 136 | 68 | 128
  QTc Fridericia: Increase from Baseline [30-60] msec | 5 | 1 | 3
  QTc Fridericia: Increase from Baseline >60 msec: number analyzed (Participants) | 136 | 68 | 128
  QTc Fridericia: Increase from Baseline >60 msec | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Physical Examination Abnormalities: Combined Stage 1 and Stage 2
Description: Physical examination included: Head, Heart, Lung, Abdomen, Musculo/Skeletal, Skin, and Mental Status. Abnormality in physical examination was based on investigator's discretion. Results are based on the treatment emergent period which was defined as time from the first IMP administration up to the last IMP administration in EFC15392 study + 30 days or up to the first visit in LTS15823 study, whichever comes earlier.
Time Frame: Baseline, Month 18, Month 24
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 200 | 78 | 199
Participants
  Baseline: Head: number analyzed (Participants) | 200 | 78 | 198
  Baseline: Head | 1 | 1 | 4
  Baseline: Heart: number analyzed (Participants) | 200 | 78 | 198
  Baseline: Heart | 2 | 1 | 1
  Baseline: Lung: number analyzed (Participants) | 200 | 78 | 198
  Baseline: Lung | 0 | 0 | 0
  Baseline: Abdomen: number analyzed (Participants) | 200 | 78 | 198
  Baseline: Abdomen | 15 | 12 | 24
  Baseline: Musculo/Skeletal: number analyzed (Participants) | 199 | 78 | 198
  Baseline: Musculo/Skeletal | 5 | 1 | 4
  Baseline: Skin: number analyzed (Participants) | 199 | 78 | 198
  Baseline: Skin | 7 | 2 | 3
  Baseline: Mental Status: number analyzed (Participants) | 200 | 78 | 198
  Baseline: Mental Status | 0 | 0 | 0
  Month 18: Head: number analyzed (Participants) | 49 | 49 | 47
  Month 18: Head | 0 | 0 | 1
  Month 18: Heart: number analyzed (Participants) | 49 | 49 | 47
  Month 18: Heart | 0 | 0 | 1
  Month 18: Lung: number analyzed (Participants) | 49 | 49 | 47
  Month 18: Lung | 0 | 0 | 0
  Month 18: Abdomen: number analyzed (Participants) | 49 | 49 | 47
  Month 18: Abdomen | 2 | 1 | 0
  Month 18: Musculo/Skeletal: number analyzed (Participants) | 49 | 49 | 47
  Month 18: Musculo/Skeletal | 0 | 0 | 1
  Month 18: Skin: number analyzed (Participants) | 49 | 49 | 47
  Month 18: Skin | 1 | 1 | 0
  Month 18: Mental Status: number analyzed (Participants) | 49 | 49 | 47
  Month 18: Mental Status | 1 | 0 | 0
  Month 24: Head: number analyzed (Participants) | 7 | 4 | 7
  Month 24: Head | 0 | 0 | 0
  Month 24: Heart: number analyzed (Participants) | 7 | 4 | 7
  Month 24: Heart | 0 | 0 | 0
  Month 24: Lung: number analyzed (Participants) | 7 | 4 | 7
  Month 24: Lung | 0 | 0 | 0
  Month 24: Abdomen: number analyzed (Participants) | 7 | 4 | 7
  Month 24: Abdomen | 0 | 0 | 0
  Month 24: Musculo/Skeletal: number analyzed (Participants) | 7 | 4 | 7
  Month 24: Musculo/Skeletal | 0 | 0 | 0
  Month 24: Skin: number analyzed (Participants) | 7 | 4 | 7
  Month 24: Skin | 0 | 0 | 0
  Month 24: Mental Status: number analyzed (Participants) | 7 | 4 | 7
  Month 24: Mental Status | 0 | 0 | 0

19. Secondary Outcome: Change From Baseline in Beck Depression Inventory-II (BDI-II) Score: Combined Stage 1 and Stage 2
Description: The Beck Depression Inventory-II (BDI-II) is a 21-item questionnaire used to assess depression. Most items are rated on a 4-point scale from 0 to 3, and a few items are rated on a 7-point scale. Individual item scores are added to get a total BDI-II score from 0 to 63. The higher the total score, the more severe the depression, and the lower the total score, the less severe the depression.
Time Frame: Baseline, Months 3, 6, 9, 12, 15, 18, 21, and 24, Last on-treatment value up to last IMP + 1 day (anytime during the maximum duration of 25 months)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 200 | 78 | 199
score on a scale
  Baseline: number analyzed (Participants) | 191 | 77 | 194
  Baseline | 4.0 (4.7) | 3.0 (4.1) | 3.4 (4.1)
  Change at Month 3: number analyzed (Participants) | 147 | 73 | 153
  Change at Month 3 | -0.1 (4.0) | 0.7 (4.0) | 0.7 (4.3)
  Change at Month 6: number analyzed (Participants) | 122 | 68 | 128
  Change at Month 6 | -0.6 (4.2) | 0.9 (4.2) | 0.3 (3.9)
  Change at Month 9: number analyzed (Participants) | 92 | 67 | 100
  Change at Month 9 | -0.3 (4.8) | 0.1 (3.7) | 0.7 (4.9)
  Change at Month 12: number analyzed (Participants) | 58 | 61 | 63
  Change at Month 12 | -1.9 (3.9) | 0.2 (4.7) | 1.5 (5.3)
  Change at Month 15: number analyzed (Participants) | 54 | 56 | 54
  Change at Month 15 | -1.5 (4.4) | -0.1 (4.4) | -0.3 (4.0)
  Change at Month 18: number analyzed (Participants) | 42 | 46 | 43
  Change at Month 18 | -1.0 (4.9) | 0.5 (3.0) | 0.0 (3.5)
  Change at Month 21: number analyzed (Participants) | 24 | 28 | 32
  Change at Month 21 | 1.0 (9.5) | -0.1 (1.3) | 1.1 (2.8)
  Change at Month 24: number analyzed (Participants) | 4 | 4 | 7
  Change at Month 24 | -0.3 (0.5) | 0.8 (2.2) | 0.3 (1.7)
  Change at Last on-treatment value: number analyzed (Participants) | 155 | 74 | 164
  Change at Last on-treatment value | -0.5 (5.1) | 0.1 (4.0) | 0.3 (4.6)

20. Secondary Outcome: Number of Participants With Worsening Lens Opacity From Baseline During the Treatment-emergent Period: Combined Stage 1 and Stage 2
Description: Worsening of lens opacity classification system (LOCS) III score or World Health Organization (WHO) grade in nuclear opacification, cortical opacification and posterior subcapsular opacification were assessed for 'Any eye', 'Unilateral' and 'Bilateral' separately. A participant could be counted in all the 3 categories. In each category, the worst case was taken into account. To be evaluable for 'Any', a participant had to have at least one eye evaluable, whereas, for 'Unilateral' and 'Bilateral', a participant had to have both eyes evaluable. Therefore, the sum of 'Unilateral' + 'Bilateral' is not necessarily equal to 'Any' in the below table. The difference observed in 'Nuclear Opacification' in 15 mg group, comes from that 1 participant who had Unilateral worsening at a given visit and a Bilateral worsening at another visit. Therefore, this participant was counted as 'Unilateral', 'Bilateral' and counted only once in 'Any'. Results are based on the TE period.
Time Frame: as for outcome 11
Population: Analysis was performed on extended Combined Stage 1 and Stage 2 safety population. Here, "number analyzed" signifies participants with available data for each specified category. Data for this OM was planned to be collected and analyzed for combined Stage 1 and Stage 2 population as pre-specified in protocol. TE period: time from first IMP administration up to the last IMP administration in EFC15392 study + 30 days or up to the first visit in LTS15823 study, whichever comes earlier.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Venglustat 8 mg | Venglustat 15 mg
Number analyzed (Participants) | 200 | 78 | 199
Participants
  Worsening of LOCS III score >= 0.5 or WHO grade >= 1.0 in nuclear opacification: Any eye: number analyzed (Participants) | 91 | 61 | 98
  Worsening of LOCS III score >= 0.5 or WHO grade >= 1.0 in nuclear opacification: Any eye | 8 | 3 | 9
  Worsening of LOCS III score >= 0.5 or WHO grade >= 1.0 in nuclear opacification: Unilateral: number analyzed (Participants) | 91 | 61 | 98
  Worsening of LOCS III score >= 0.5 or WHO grade >= 1.0 in nuclear opacification: Unilateral | 0 | 0 | 4
  Worsening of LOCS III score >= 0.5 or WHO grade >= 1.0 in nuclear opacification: Bilateral: number analyzed (Participants) | 91 | 61 | 98
  Worsening of LOCS III score >= 0.5 or WHO grade >= 1.0 in nuclear opacification: Bilateral | 8 | 3 | 6
  Worsening of LOCS III score >= 0.8 or WHO grade >= 1.0 in cortical opacification: Any eye: number analyzed (Participants) | 84 | 61 | 87
  Worsening of LOCS III score >= 0.8 or WHO grade >= 1.0 in cortical opacification: Any eye | 4 | 4 | 4
  Worsening of LOCS III score >= 0.8 or WHO grade >= 1.0 in cortical opacification: Unilateral: number analyzed (Participants) | 83 | 61 | 87
  Worsening of LOCS III score >= 0.8 or WHO grade >= 1.0 in cortical opacification: Unilateral | 1 | 0 | 1
  Worsening of LOCS III score >= 0.8 or WHO grade >= 1.0 in cortical opacification: Bilateral: number analyzed (Participants) | 83 | 61 | 87
  Worsening of LOCS III score >= 0.8 or WHO grade >= 1.0 in cortical opacification: Bilateral | 2 | 4 | 3
  Worsening of LOCS III score>=0.5 or WHO grade >= 1.0 in posterior subcapsular opacification:Any eye: number analyzed (Participants) | 81 | 56 | 87
  Worsening of LOCS III score>=0.5 or WHO grade >= 1.0 in posterior subcapsular opacification:Any eye | 2 | 2 | 3
  Worsening of LOCS III score>=0.5 or WHO grade >=1.0 in posterior subcapsularopacification:Unilateral: number analyzed (Participants) | 81 | 56 | 87
  Worsening of LOCS III score>=0.5 or WHO grade >=1.0 in posterior subcapsularopacification:Unilateral | 0 | 1 | 1
  Worsening of LOCS III score>=0.5 or WHO grade >=1.0 in posterior subcapsular opacification:Bilateral: number analyzed (Participants) | 81 | 56 | 87
  Worsening of LOCS III score>=0.5 or WHO grade >=1.0 in posterior subcapsular opacification:Bilateral | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: From the first IMP administration up to the last IMP administration in EFC15392 study + 30 days (i.e., up to 25 months) or up to the first visit in LTS15823 study, whichever comes earlier
Description: Reported AEs were TEAEs that developed/worsened in grade or became serious during TE period (time from the first IMP administration up to the last IMP administration in EFC15392 study + 30 days or up to the first visit in LTS15823 study, whichever comes earlier). Analysis was performed on the Stage 1 and Stage 2 safety population.
Arm/Group | Stage 1- Placebo | Stage 1- Venglustat 8 mg | Stage 1- Venglustat 15 mg | Stage 2- Placebo | Stage 2- Venglustat 15 mg
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/78 | 0/80 | 0/122 | 0/119
Serious Adverse Events (participants affected / at risk) | 8/78 | 15/78 | 19/80 | 6/122 | 7/119
Other Adverse Events (participants affected / at risk) | 42/78 | 46/78 | 48/80 | 32/122 | 48/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1- Placebo (N=78) | Stage 1- Venglustat 8 mg (N=78) | Stage 1- Venglustat 15 mg (N=80) | Stage 2- Placebo (N=122) | Stage 2- Venglustat 15 mg (N=119)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected Cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Cyst Infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mediastinum Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial Aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental Cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large Intestinal Stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Renal Cyst Haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal Cyst Ruptured (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal Haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic Cyst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaw Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1- Placebo (N=78) | Stage 1- Venglustat 8 mg (N=78) | Stage 1- Venglustat 15 mg (N=80) | Stage 2- Placebo (N=122) | Stage 2- Venglustat 15 mg (N=119)
Covid-19 (Infections and infestations) | 5 (5) | 6 (6) | 1 (1) | 3 (3) | 7 (7)
Conjunctivitis (Infections and infestations) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (13) | 5 (5) | 6 (9) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 4 (4) | 6 (8) | 4 (4) | 6 (7)
Urinary Tract Infection (Infections and infestations) | 6 (6) | 5 (6) | 7 (15) | 3 (4) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4) | 4 (4) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 6 (6) | 8 (9) | 11 (14) | 7 (8) | 8 (8)
Cataract Cortical (Eye disorders) | 5 (5) | 2 (4) | 3 (3) | 1 (1) | 2 (2)
Cataract Nuclear (Eye disorders) | 5 (5) | 2 (2) | 3 (4) | 1 (1) | 2 (2)
Dry Eye (Eye disorders) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 5 (5) | 7 (7) | 4 (4) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (8) | 8 (8) | 1 (1) | 7 (8)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 6 (6) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (6) | 7 (9) | 0 (0) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 6 (7) | 8 (8) | 5 (5) | 2 (2)
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 4 (5) | 0 (0) | 4 (5) | 2 (2)
Fatigue (General disorders) | 1 (1) | 4 (5) | 9 (9) | 3 (3) | 2 (2)
Influenza Like Illness (General disorders) | 1 (1) | 5 (5) | 1 (1) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Following decision to discontinue EFC15392 based on the futility analysis, the two-steps analysis initially planned were not applicable, therefore only the final analysis of all safety endpoints (laboratory, vital sign, ECG, physical examination, BDI-II, and lens opacity) were performed on extended combined Stage 1 and Stage 2 safety population only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT03523728/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT03523728/SAP_001.pdf